CLINICAL TRIAL: NCT04137120
Title: Assessment of the Safety and Drug Utilization of Intravitreal Aflibercept Injection in Mexican Routine Clinical Practice for the Treatment of Wet Age Related Macular Degeneration (wAMD), Diabetic Macular Edema (DME), Macular Edema Secondary to Central Retinal Vein Occlusion (CRVO), Macular Edema Secondary to Branch Retinal Vein Occlusion (BRVO) and Myopic Neovascularization (mCNV). A Post-authorization Safety Study (PASS).
Brief Title: Study to Gather Information on the Safety and Use of Aflibercept Injections Into the Eye for the Treatment of Eye Disorders in Mexican Routine Clinical Practice
Acronym: MAIA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19212
Record Dates: First submitted 2019-10-22; First posted 2019-10-23 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Retinal Disease
Keywords: Aflibercept; Intravitreal injection; Ocular disease; Wet age-related macular degeneration (wAMD); Diabetic macular edema (DME); Macular edema secondary to central retinal vein occlusion (CRVO); Macular edema secondary to branch retinal vein occlusion (BRVO); Myopic choroidal neovascularization (mCNV); Mexico
MeSH Terms: conditions — Retinal Diseases | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients_Ocular disease: Adult patients treated for wet age-related macular degeneration (wAMD), or diabetic macular edema (DME), or macular edema secondary to central retinal vein occlusion (CRVO), or macular edema secondary to branch retinal vein occlusion (BRVO) or myopic choroidal neovascularization (mCNV) in routine clinical practice in Mexico (overall cohort)
  Interventions: Drug: Aflibercept (BAY86-5321, Eylea)

INTERVENTIONS:
Drug: Aflibercept (BAY86-5321, Eylea) — Intravitreal injection of aflibercept as scheduled by treating physician
  Other Names: Eylea®; Eylia®; Wetlia®; VEGF Trap-Eye

SUMMARY:
The study aims to collect data on the safety and use of intravitreal aflibercept injections into the eye for the treatment of eye disorders that cause blurred vision or a blind spot due to abnormal or blocked blood vessels. Data will be collected from patients who are being treated for such eye disorders in Mexican routine clinical practice.

DETAILED DESCRIPTION:
The primary objective is to assess the safety of intravitreal aflibercept injections in patients with wet age-related macular degeneration (wAMD), myopic choroidal neovascularization (mCNV), diabetic macular edema (DME), macular edema secondary to central retinal vein occlusion (CRVO) or macular edema secondary to branch retinal vein occlusion (BRVO).

Secondary objectives comprise the comparison of the aflibercept safety profile between defined subgroups and the assessment of the real-world application of intravitreal aflibercept injections with special focus on CRVO, BRVO and mCNV indications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of a wet age-related macular degeneration (wAMD), diffuse diabetic macular edema (DME), macular edema secondary to central retinal vein occlusion (CRVO), macular edema secondary to branch retinal vein occlusion (BRVO) or myopic choroidal neovascularization (mCNV);
* Decision to initiate treatment with intravitreal aflibercept was made as per investigator's routine treatment practice and independently of study inclusion;
* Treatment naïve or pre-treated for macular diseases (to anti-VEGF and steroid intravitreal treatments); patients who underwent laser photocoagulation and/or are being treated with panretinal photocoagulation therapies are eligible for study participation;
* If of childbearing potential, female willing to use effective contraception during treatment and for at least 3 months after the last intravitreal injection of aflibercept

Exclusion Criteria:

* Patient diagnosed with two or more of the studied indications in the same eye (wAMD, DME, CRVO, BRVO and mCNV);
* Patients that were already treated with anti-VEGF or steroids are allowed to be enrolled only if they received the last dose of anti-VEGF 3 or more months ago and in the case of a steroid implant 6 months after the last dose;
* Current treatment with other intravitreal therapies
* Contra-indications according to Eylea's / Wetlia's local marketing authorization:

  * Ocular or periocular infection
  * Active intraocular Inflammation
  * Known hypersensitivity to aflibercept or to any of its excipients
  * Pregnant or lactating women.
* Participation in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with macular disease in Mexican routine practice
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Number of ocular adverse events | Up to 12 months
Number of serious ocular adverse events | Up to 12 months
Seriousness reason for ocular adverse events | Up to 12 months
  Seriousness reasons may be death, life-threatening character of event, hospitalization or prolongation of hospitalization, congenital anomaly/ birth defect, persistent or significant impairment, or medical relevance of adverse event.
Severity of ocular adverse events | Up to 12 months
  The severity of adverse events is classified as mild, moderate or severe by treating physician.
Number of treatment-related ocular adverse events | Up to 12 months
Number of injection-related ocular adverse events | Up to 12 months
Action taken with drug after ocular adverse event | Up to 12 months
  Options: Withdrawn, Interrupted, Injection schedule changed, Injection schedule not changed
Clinical outcome of ocular adverse event | Up to 12 months
  Options: Resolved, Resolving, Resolved with sequelae, Not resolved, Fatal, Unknown
Duration of ocular adverse events | Up to 12 months
Duration of patient follow-up after ocular adverse event (in months) | Up to 12 months
Number of non-ocular adverse events | Up to 12 months
Number of serious non-ocular adverse events | Up to 12 months
Seriousness reason for non-ocular adverse events | Up to 12 months
  Seriousness reasons may be death, life-threatening character of event, hospitalization or prolongation of hospitalization, congenital anomaly/ birth defect, persistent or significant impairment, or medical relevance of adverse event.
Severity of non-ocular adverse events | Up to 12 months
  The severity of adverse events is classified as mild, moderate or severe by treating physician.
Number of treatment-related non-ocular adverse events | Up to 12 months
Number of injection-related non-ocular adverse events | Up to 12 months
Action taken with drug after non-ocular adverse event | Up to 12 months
  Options: Withdrawn, Interrupted, Injection schedule changed, Injection schedule not changed
Clinical outcome of non-ocular adverse event | Up to 12 months
  Options: Resolved, Resolving, Resolved with sequelae, Not resolved, Fatal, Unknown
Duration of non-ocular adverse events | Up to 12 months
Duration of patient follow-up after non-ocular adverse event (in months) | Up to 12 months

SECONDARY OUTCOMES:
Total number of injections with intravitreal aflibercept per study eye | Up to 12 months
Time between injections in the study eye (in days) | Up to 12 months
Time between injections in the study eye and fellow eye (in days) | Up to 12 months
Number of patients receiving bilateral treatment | Up to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.